CLINICAL TRIAL: NCT04130217
Title: Ultrasonographic Evaluation of the Effect of Recruitment Maneuvers and Positive End-expiratory Pressure on Diaphragmatic Functions and Atelectasis in Obese Patients Undergoing Laparoscopic Sleeve Gastrectomy: A Randomized Controlled Study
Brief Title: Ultrasonograpahic Evaluation of Diaphragmatic Functions in Obese Patients Undergoing Laparoscopic Sleeve Gastrectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Shereen Elsayed Abd Ellatif, lecturer of anesthesia and surgical intensive care, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 5610/20-1-2019
Record Dates: First submitted 2019-10-14; First posted 2019-10-17 (Actual); Last update posted 2020-06-26 (Actual); Status verified 2020-06

CONDITIONS: Bariatric Surgery Candidate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (No Intervention): patients will be intraoperatively mechanically ventilated without PEEP nor RM.
- PEEP Group (Experimental): patients will be intraoperatively mechanically ventilated with PEEP of 5 cmH2O.
  Interventions: Procedure: addition of positive end expiratory pressure in ventilated patients
- PEEP and RM Group (Experimental): patients will be intraoperatively mechanically ventilated with PEEP of 5 cmH2O and intermittent four times of RM consisting of maintaining airway pressure 40 cmH2O for 40 sec.
  Interventions: Procedure: addition of positive end expiratory pressure and recruitment maneuver in ventilated patients

INTERVENTIONS:
Procedure: addition of positive end expiratory pressure in ventilated patients — patients will be intraoperatively mechanically ventilated with PEEP of 5 cmH2O.
  Arms: PEEP Group
Procedure: addition of positive end expiratory pressure and recruitment maneuver in ventilated patients — patients will be intraoperatively mechanically ventilated with PEEP of 5 cmH2O and intermittent four times of RM consisting of maintaining airway pressure 40 cmH2O for 40 sec.
  Arms: PEEP and RM Group

SUMMARY:
Major laparoscopic sleeve gastrectomy surgery requires steep Trendelenburg position with pneumoperitoneum for a long time leading to decrease pulmonary compliance and lung volumes due to cephalic displacement and decrease excursion of the diaphragm, consequently leading to the possibility of atelectasis formation. Different strategies have been proposed to reduce atelectasis and other pulmonary complications in obese patients as induction of anesthesia in the head up position with or without CPAP, protective intraoperative mechanical ventilation with high or low levels of PEEP and implementation of Recruitment Maneuvers. Up to investigators' knowledge, there is no study done to evaluate the effect of intraoperative use of PEEP and alveolar recruitment maneuver on diaphragmatic function and incidence of atelectasis via ultrasonography in obese patients undergoing laparoscopic sleeve gastrectomy.

DETAILED DESCRIPTION:
Bariatric surgery is one of the fastest-growing areas of surgery. It is the most effective treatment for morbid obesity and its secondary co-morbidities. Although there is no gold standard surgical procedure for obesity management, laparoscopic sleeve gastrectomy (LSG) is considered to be the first choice procedure and recently it becomes the most common bariatric surgical procedure performed worldwide. LSG is preferred to open techniques because it is associated with less incisional pain, shorter operative time, fewer pulmonary complications, and earlier hospital discharge.

However, laparoscopic procedures are operated under general anesthesia that decreases functional residual capacity (FRC) and enhances atelectasis. Also, it is performed in conjunction with intra-abdominal CO2 insufflation and subsequent increase in the intra-abdominal pressure, this CO2 pneumoperitoneum together with the steep Trendelenburg position which is maintained for long period in LSG, result in cephalic displacement of the diaphragm leading to several respiratory changes as decreased FRC and vital capacity (VC), decrease pulmonary compliance, consequently resulting in atelectasis formation in the dependent lung regions. Moreover, obese patients are more prone to develop peri-operative atelectasis and postoperative pulmonary complications that are almost twice the risk among healthy subjects.

This alteration in FRC and lung volumes are more clinically relevant as it can result in small airway closure and further ventilation-perfusion mismatch that may lead to postoperative hypoxemia and respiratory complications. Several studies revealed that these lung volumes decrease and its ensuing complications are not only due to cephalic displacement of the diaphragm but also due to decreased diaphragmatic excursion.

Several strategies have been proposed to reduce the incidence of atelectasis and other pulmonary complications such as induction of anesthesia in the head-up position with or without a continuous positive airway pressure (CPAP), use of intraoperative PEEP and implementation of alveolar recruitment maneuver (RM) but it seems that the latter may be an effective method according to several studies conducted on morbidly obese patients undergoing laparoscopic surgery and demonstrated that intraoperative recruitment of lung volume improves the respiratory mechanics and oxygenation. While other studies showed that the application of PEEP intraoperatively during laparoscopic colorectal surgery is helpful for preserving diaphragmatic excursion and consequently reduce the incidence of atelectasis.

It is worth mentioning that ultrasonography (US) can play an important role in evaluating the diaphragmatic structure by measuring diaphragmatic thickness as well as diaphragmatic function by measuring diaphragmatic excursion/displacement (DD). It is a promising bedside test to evaluate the structure and dynamic function of diaphragm peri-operatively and in critically ill patients to predict the expected outcome.

The investigators hypothesize that performing RM in addition to PEEP may have an impact on improving diaphragmatic function in terms of diaphragmatic excursion evaluated by ultrasonography in obese patients undergoing LSG. Therefore; it may decrease the incidence of postoperative pulmonary complications.

ELIGIBILITY:
Inclusion Criteria:

* Patient acceptance.
* Age 21-60 years old.
* BMI ≥35 kg/m2
* ASA II and ASA III.
* Elective laparoscopic sleeve gastrectomy under general anesthesia.

Exclusion Criteria:

* Preoperative diagnosis of obstructive sleep apnea by using the STOP-BANG questionnaire (Snoring, Tiredness during the daytime, observed apnea, high blood pressure, Body mass index over 35, Age, Neck circumference, and Gender)
* History of pneumothorax or right-side heart failure.
* History of chronic respiratory disease, diaphragmatic disease, or neuromuscular disease.
* Any contraindication for laparoscopic surgery or head-down position.
* Any history with post esophageal or thoracic surgeries due to intraoperative diaphragmatic manipulation.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 69 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-02-01 (Actual)

PRIMARY OUTCOMES:
changes of Diaphragmatic excursion (DD) | 24 hour postoperative
  will be measured by low frequency probe of Sonosite M Turbo ultrasonography, measurements will be taken before induction of anaesthesia, 5 min after completion of pneumoperitoneum, 5 min after adopting Trendelenburg position, 60 min later with pneumoperitoneum and Trendelenburg position, 5 min after exsufflation of pneumoperitoneum and patient placed back in the supine position, 15 min after arrival of patient in the recovery room and 24h postoperatively.

SECONDARY OUTCOMES:
Incidence of lung atelectasis | 24 hour postoperative
  atelectasis will be assessed by a linear probe of Sonosite M Turbo ultrasonography. Its measurements will be taken just before induction of anaesthesia, 15 min after arrival of the patient in the recovery room and 24h postoperatively.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of medicine, zagazig university, Zagazig, Elsharqya, Egypt

IPD SHARING:
Plan to Share IPD: Yes
planned after the completion of the study and publication
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: after the publication of the study
Access Criteria: contact of principal investigator

REFERENCES:
- [Background] Felsenreich DM, Prager G, Kefurt R, Eilenberg M, Jedamzik J, Beckerhinn P, Bichler C, Sperker C, Krebs M, Langer FB. Quality of Life 10 Years after Sleeve Gastrectomy: A Multicenter Study. Obes Facts. 2019;12(2):157-166. doi: 10.1159/000496296. Epub 2019 Mar 15. PMID 30879011
- [Background] Guetta O, Vakhrushev A, Dukhno O, Ovnat A, Sebbag G. New results on the safety of laparoscopic sleeve gastrectomy bariatric procedure for type 2 diabetes patients. World J Diabetes. 2019 Feb 15;10(2):78-86. doi: 10.4239/wjd.v10.i2.78. PMID 30788045
- [Background] 3- Sarandan M, Guragata-Balasa C, Papurica M, Duta C, Hordovan E, Rus C, et al. Anesthesia in laparoscopic bariatric surgery (gastric sleeve) - preliminary experience. TMJ 2011; 61(1): 26-31.
- [Background] Reinius H, Jonsson L, Gustafsson S, Sundbom M, Duvernoy O, Pelosi P, Hedenstierna G, Freden F. Prevention of atelectasis in morbidly obese patients during general anesthesia and paralysis: a computerized tomography study. Anesthesiology. 2009 Nov;111(5):979-87. doi: 10.1097/ALN.0b013e3181b87edb. PMID 19809292
- [Background] Suh MK, Seong KW, Jung SH, Kim SS. The effect of pneumoperitoneum and Trendelenburg position on respiratory mechanics during pelviscopic surgery. Korean J Anesthesiol. 2010 Nov;59(5):329-34. doi: 10.4097/kjae.2010.59.5.329. Epub 2010 Nov 25. PMID 21179295
- [Background] 6- Rashwan DAE, Mahmoud HE, Nofal WH, Sabek EA. Ultrasonographic Evaluation of the Effect of Positive End-expiratory Pressure on Diaphragmatic Functions in Patients Undergoing Laparoscopic Colorectal Surgery: A Prospective Randomized Comparative Study. J Anesth Clin Res. 2018; 9(7): 843-51.
- [Background] Matamis D, Soilemezi E, Tsagourias M, Akoumianaki E, Dimassi S, Boroli F, Richard JC, Brochard L. Sonographic evaluation of the diaphragm in critically ill patients. Technique and clinical applications. Intensive Care Med. 2013 May;39(5):801-10. doi: 10.1007/s00134-013-2823-1. Epub 2013 Jan 24. PMID 23344830